CLINICAL TRIAL: NCT01887145
Title: Endoscopic Versus Open Carpal Tunnel Release: 10 to 15 Years Follow-up of a Randomized Controlled Trial
Brief Title: Comparison of Long-term Outcomes Following Endoscopic or Open Surgery for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLM-CTSRCT-2
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; Surgery; Outcomes
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Endoscopy; Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open surgery (Active Comparator): Open surgery is Open carpal tunnel release
  Interventions: Procedure: Open surgery
- Endoscopic surgery (Experimental): Endoscopic surgery is 2-portal endoscopic carpal tunnel release
  Interventions: Procedure: Endoscopic surgery

INTERVENTIONS:
Procedure: Endoscopic surgery — Surgery dwas done under local anesthesia injected at the portal sites only. Tourniquet was used. Each of the two skin incisions in the endoscopic procedure was 1 cm long. With the endoscope inserted from the distal portal and a hook knife inserted from the proximal portal, the transverse carpal ligament was divided from its distal edge to its proximal edge. Incisions were closed with non-absorbables sutures and a soft dressing was applied. Sutures were removed 10 days postoperatively.
  Other Names: Endoscopic carpal tunnel release surgery
  Arms: Endoscopic surgery
Procedure: Open surgery — Open carpal tunnel release using conventional open technique under local anesthesia and tourniquet. The incision in the open procedure extended from about 1 cm proximal to 3 cm distal to the wrist crease. The transverse carpal ligament was divided; no additional procedures were performed. a soft dressing was applied. Dressing and sutures were removed 10 days postoperatively.
  Other Names: Open carpal tunnel release surgery
  Arms: Open surgery

SUMMARY:
No randomized trials have compared long-term outcomes following endoscopic and open carpal tunnel release in patients with carpal tunnel syndrome (CTS). The investigators conducted a single-center randomized controlled trial between January 1998 and December 2002, including 128 patients (25 to 60 years) with clinically diagnosed and electrophysiologically confirmed idiopathic CTS. The outcome measures included the validated CTS symptom severity and functional status scales completed at baseline and 1 year postoperatively. The trial showed that the 1-year outcomes of open and endoscopic carpal tunnel release regarding symptoms and function were equivalent. This extended follow-up of the randomized trial will primarily measure the symptom outcomes at 10-15 years after surgery. A questionnaire will be sent by mail to the patients. The questionnaire will consist of the CTS symptom severity and functional status scales, the 6-item CTS symptoms scale (CTS-6), the 11-item disabilities of the arm, shoulder and hand (QuickDASH), the 2-item palmar pain scale, and a visual analog scale about treatment satisfaction. The patients will also be asked about whether they had undergone further surgery for CTS in the same or contralateral hand after their operation in the randomized trial. The completed questionnaires will be scanned into a database. The scores for the different scales will be calculated. Analysis will include comparison between the open and endoscopic groups as well as within-group changes of scores from 1 year to 10-15 years.

ELIGIBILITY:
Inclusion Criteria (original trial):

* Primary idiopathic carpal tunnel syndrome
* age 25-60 years
* currently employed
* duration of symptoms of at least three months
* inadequate response to six weeks' treatment with wrist splint
* symptoms of classic or probable carpal tunnel syndrome according to the diagnostic criteria in the Katz hand diagram, and nerve conduction test showing median neuropathy at the wrist (distal motor latency ≥4.5 milliseconds, wrist-digit sensory latency ≥3.5 milliseconds, or sensory conduction velocity at the carpal tunnel segment <40 metres/second but no other abnormalities.

Exclusion Criteria (original trial):

Inflammatory joint disease

* diabetes mellitus, thyroid disorder, pregnancy, trauma to the affected hand during the preceding year
* previous carpal tunnel release surgery in the affected hand
* carpal tunnel release surgery in the contralateral hand during the preceding year
* symptoms of carpal tunnel syndrome in the contralateral hand not adequately relieved by splint at the time of enrollment
* current sick leave because of disorders other than carpal tunnel syndrome
* inability to complete questionnaires because of language problem or cognitive disorder.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in CTS symptom severity score | Baseline to 10-15 years postoperatively

SECONDARY OUTCOMES:
Rate of repeat surgery | 10-15 years postoperatively
Change in CTS functional status score | from baseline and 1 year to 10-15 years postoperatively
Residual pain in the scar or proximal palm | 10-15 years postoperatively
Patient satisfaction with the results of surgery | 10-15 years postoperatively
Change in CTS symptom severity score | 1 year to 10-15 years postoperatively

OTHER OUTCOMES:
CTS-6 score | 10-15 years postoperatively
QuickDASH score | 10-15 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Isam Atroshi, MD, PhD, Principal Investigator — Clinical Sciences, Lund University, Sweden

REFERENCES:
- [Background] Atroshi I, Larsson GU, Ornstein E, Hofer M, Johnsson R, Ranstam J. Outcomes of endoscopic surgery compared with open surgery for carpal tunnel syndrome among employed patients: randomised controlled trial. BMJ. 2006 Jun 24;332(7556):1473. doi: 10.1136/bmj.38863.632789.1F. Epub 2006 Jun 15. PMID 16777857
- [Derived] Atroshi I, Hofer M, Larsson GU, Ranstam J. Extended Follow-up of a Randomized Clinical Trial of Open vs Endoscopic Release Surgery for Carpal Tunnel Syndrome. JAMA. 2015 Oct 6;314(13):1399-401. doi: 10.1001/jama.2015.12208. No abstract available. PMID 26441187